CLINICAL TRIAL: NCT00313053
Title: A Phase I Study of mAb 216 With Chemotherapy for the Treatment of Pediatric Patients With Relapsed or Refractory B-progenitor Acute Lymphoblastic Leukemia
Brief Title: Study of mAb 216 With Chemotherapy for Treatment of Pediatric Relapsed or Refractory B-progenitor Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Clare Twist (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Clare Twist, Associate Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDSMAB216; 95343; CA85199-01; NCT00313053; PEDSMAB216; 13822 (Other: Stanford IRB)
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2012-11

CONDITIONS: Leukemia, Lymphocytic, Acute; Leukemia; Acute Lymphoid Leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Vincristine

ARMS (1):
- Human mAb 216 (Experimental)
  Interventions: Drug: Human mAb 216; Drug: Vincristine

INTERVENTIONS:
Drug: Human mAb 216 — Two treatment courses of mAb infusion will be given, with the same dose of antibody administered on Day 0 and on Day 7.
Drug: Vincristine — Vincristine 1.5 mg/m2/dose (max dose = 2 mg) IVP on weekly x 4 doses (Days 7, 14, 21, 28)

SUMMARY:
This is a phase I trial in patients with relapsed or refractory leukemia of a human monoclonal antibody that kills B cell acute lymphoblastic leukemia. The trial will study the safety, pharmacokinetics, and anti-tumor activity of the antibody given as a single agent and with vincristine.

ELIGIBILITY:
Inclusion Criteria:- Patients must be > than 12 months at the time of study entry.

* Patients must have had histologic verification of B-lineage ALL with bone marrow relapse or refractory disease that is unresponsive to traditional chemotherapy.
* For patients WITHOUT prior allogeneic bone marrow transplant (BMT):

  * Second or subsequent bone marrow relapse
  * Primary refractory marrow disease
  * M3 marrow (> 25% blasts)
* For patients WITH prior allogeneic BMT:

  * First or subsequent bone marrow relapse post-BMT
  * M3 marrow or M2 (> 5% and < 25% blasts) if cytogenetic or variable number tandem repeat (VNTR) confirmation
* Confirmation of antibody reactivity
* Patient's leukemic blasts (peripheral blood or marrow) must be documented to bind mAb 216 in vitro (Teng lab).
* Patient's red blood cell (RBC) documented to NOT express fetal "i" antigen and RBC shown to NOT bind mAb 216 in vitro (Teng lab)
* Patient must not be eligible for therapies of higher priority
* Performance level Karnofsky 50% for patients > 10 years of age and Lansky >= 50 for patients <= 10 years of age.
* Life expectancy must be at least 8 weeks.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study:

  * Myelosuppressive chemotherapy: must not have been received within 2 weeks of entry onto this study.
  * Biologic: at least 7 days since the completion of therapy with a biologic agent.
* No hematologic criteria for white blood cell (WBC), hemoglobin (Hgb), or platelets
* Patients with thrombocytopenia should be responsive to platelet transfusions and must not have uncontrolled bleeding.
* Adequate renal function defined as: a serum creatinine that is less than or equal to 1.5 x normal for age
* Adequate liver function defined as: total bilirubin <= 1.5 x upper limit of normal (ULN) for age, and SGPT (ALT) <= 5 x upper limit of normal (ULN) for age
* Adequate cardiac function defined as: shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study.
* All patients and/or their parents or legal guardians must sign a written informed consent/assent.
* All Institutional Review Board (IRB) and Food and Drug Administration (FDA) requirements for human studies must be met. Exclusion Criteria:- Central nervous system (CNS) 3 or refractory CNS leukemia
* Isolated extramedullary relapse
* Uncontrolled infection
* Lack of mAb 216 binding to patient's leukemic blasts in vitro
* Binding of mAb 216 to the"i" antigen on patient's erythrocytes
* Prior treatment with rituximab

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2004-09; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose without toxicity
Safety

SECONDARY OUTCOMES:
Decrease in leukemic blasts

CONTACTS AND LOCATIONS:
Overall Officials: Clare J. Twist M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States